CLINICAL TRIAL: NCT02575118
Title: Concentration of Bisphenol A in Saliva and Urine Before and After Treatment With Polymer-based Dental Filling Materials
Brief Title: Bisphenol A in Saliva and Urine Related to Placement of Dental Composites
Status: Completed | Type: Observational
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Hordaland County (Other Government)
Responsible Party: Sponsor
Other Study IDs: REK 2014/1529
Record Dates: First submitted 2015-10-05; First posted 2015-10-14 (Estimated); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2018-05

CONDITIONS: Dental Polymer Based Filling Material

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva Urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Restoration of dental caries with dental composite

SUMMARY:
It has been reported that therapy with polymer-based dental filling materials was associated with higher concentrations of bisphenol A in saliva and urine directly after the treatment. The objective of the present project is to gain knowledge about the concentration of bisphenol A in saliva and urine before and after treatment with polymer-based dental filling materials, using sensitive analytical methods.

DETAILED DESCRIPTION:
Bisphenol A (BPA) is a xenoestrogen which has been shown to cause abnormalities in sexual development and may lead to reproductive damage in animals. In epidemiological studies BPA has been associated with various health effects. The majority of dental plastic filling materials contain polymers synthesized from BPA. Whether BPA is released in vivo from polymer-based fillings and - if so, in what doses - is not sufficiently examined. Patients scheduled for regular dental examination at the public dental clinic, Bergen Downtown District, who needs therapy with dental polymer-based filling materials and is suitable for study (inclusion / exclusion criteria) will be informed about the project. If the patient wants to participate in the study, he/she will be given written information about the study and a consent form. It is emphasized that participation in the study is voluntary and the patient will have the opportunity to read the information at home, before the next appointment at the clinic. The clinical treatment of the carious lesion(s) will be performed according to standardized procedures and materials used at the clinic. After curing, the filling will be polished according to the standard procedures. The curing lamp will be controlled and documented weekly during the project period. All treatment sessions will be scheduled in the morning before 9 am. Questions regarding food intake and dental hygiene habits will be included in questionnaires answered during the study. Samples of saliva and urine will be collected immediately before filling placement and 1 hour, 24 hours and 1 week after treatment. A saliva sample will also be collected immediately after treatment. No food or drink intake is allowed after midnight before sample collection. Only tapped water is permitted. The sampling procedure will be controlled in advance, so that the risk of contamination of samples is minimized. After collection samples will be refrigerated and stored frozen at -80 °C until analysis. Bisphenol A in saliva and urine will be determined by liquid chromatography and mass spectrometry (LC-MS). The detection limit of the method is estimated at 0.1 ng BPA/ml. The study is approved by the Regional Committee for Medical and Health Research (reference number 2014/1529). Patients who participate in the project will have to collect saliva samples five times and urine samples four times, which involves extra visits to the clinic. The biomedical outcomes (concentration of bisphenol A in saliva and urine) will be assessed in a pre-defined group of individuals. The participants may be enrolled in the study if they fulfil the criteria (including need of a dental filling). The participants do not receive the intervention (placement of a dental filling) because they are enrolled in the study. Subjects in the study will receive the therapeutic intervention, but the investigator does not assign the intervention to the subjects of the study. Thus, the study may be described as an observational study.

ELIGIBILITY:
Inclusion Criteria:

* Need for filling therapy that involves at least two surfaces with a polymer-based filling material
* Healthy patient without any chronic diseases
* Age 16 - 40 years
* Informed consent given

Exclusion Criteria:

* Drug abuse
* Smoking
* Use of snuff
* Use of dental splint
* Work at a dental clinic

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients scheduled for regular dental examination at the public dental clinic (Bergen Downtown District) and the Dental Clinic of the Student Welfare Organization in Bergen, who are in need for treatment with dental polymer-based filling materials, are suitable for study (inclusion / exclusion criteria) and have given their written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Björkman, DDS, PhD, Study Chair — NORCE Norwegian Research Centre AS
Locations (1):
- Public dental clinic, Bergen Downtown District AND Dental Clinic of the Student Welfare Organization in Bergen, Bergen, Norway

REFERENCES:
- [Result] Berge TLL, Lygre GB, Lie SA, Lindh CH, Bjorkman L. Bisphenol A in human saliva and urine before and after treatment with dental polymer-based restorative materials. Eur J Oral Sci. 2019 Oct;127(5):435-444. doi: 10.1111/eos.12647. Epub 2019 Aug 8. PMID 31392814

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Patients in need of at least one dental restoration, involving two or more tooth surfaces, with a polymer-based restorative material were informed about the study by their dental hygienist or dentist at their regular dental examination at two public dental clinics in Bergen, Norway.
Period: Overall Study
Arm/Group | Treatment Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.4 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 20
Education [Mean (Standard Deviation); unit: years] | 13.8 (1.8)
Job handling receipts [Number; unit: Number of Participants Handling Receipts] | 5

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Bisphenol A in Saliva
Description: Estimated bisphenol A (BPA) concentration (ng ml-1) in saliva
Time Frame: 1 week
Population: n=19 at 1 week follow up (since mixed effects models were used all available data, also data for participants with missing observations at some time points, were included in the model [see: Rabe-Hesketh and Skrondal. Multilevel and Longitudinal Modeling Using Stata, Volume I, Third Edition. 2012, page 279])
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
ng/ml | 0.25 [0.17 to 0.33]
Statistical Analysis 1: Comparison: Treatment Group; In one saliva sample collected before treatment, the BPA concentration was more than 100 times higher (11.6 ng/ml) than the mean value and more than 100 SD from the mean of the remaining 19 samples. This saliva sample was excluded from the statistical analysis because it was probably contaminated. One participant had breakfast before the sample time point 1 wk after treatment, and thus the samples collected from this participant at this time point were not included in the statistical analysis; Test type: Other; p < 0.05, linear mixed-effects regression models; All available data, and hence data for participants with missing observations at some time points, were included in the model; We used mixed effects models and all available data (also data for participants with missing observations at some time points) were included in the model. Using mixed effects models is a recognized method when there are missing data. Thus, data from all 20 individuals were used for estimations at all time points (see: Rabe-Hesketh and Skrondal. Multilevel and Longitudinal Modeling Using Stata, Volume I, Third Edition. 2012, page 279)

2. Primary Outcome: Concentration of Bisphenol A in Urine
Description: Estimated bisphenol A (BPA) concentration (ng ml-1) in urine
Time Frame: 1 week
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
ng/ml | 1.99 [0.97 to 3.00]
Statistical Analysis 1: Comparison: Treatment Group; One participant had breakfast before the sample time point 1 wk after treatment, and thus the samples collected from this participant at this time point were not included in the statistical analysis; Test type: Other; p < 0.05, linear mixed-effects regression models; [statistical method as in outcome 1, analysis 1]; We used mixed effects models and all available data (also data for participants with missing observations at some time points), were included in the model. Using mixed effects models is a recognized method when there are missing data. Thus, data from all 20 individuals were used for estimations at all time points (see: Rabe-Hesketh and Skrondal. Multilevel and Longitudinal Modeling Using Stata, Volume I, Third Edition. 2012, page 279)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT02575118/Prot_SAP_000.pdf